CLINICAL TRIAL: NCT04169061
Title: A Multicenter, Open-label Study to Assess the Efficacy and Safety of Acthar® Gel in Subjects With Severe Keratitis
Brief Title: Impact of Acthar on Everyday Life of Participants With Severe Keratitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNK14084113
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Keratitis
Keywords: Severe or recalcitrant keratitis
MeSH Terms: conditions — Keratitis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): Participants receive:
  * a shot of Acthar (80 units) under the skin twice a week for 12 weeks
  * a shot of Acthar (40 units) twice a week for 2 weeks
  * a shot of Acthar (40 units) once a week for 2 more weeks
  At each visit they will have medical tests and answer questions about their symptoms.
  Interventions: Drug: Acthar

INTERVENTIONS:
Drug: Acthar — Acthar gel for subcutaneous injection
  Other Names: Acthar Gel

SUMMARY:
We will need about 36 participants for this study.

Volunteers might be able to participate if:

* they have bad noninfectious keratitis
* early treatments failed or were not well tolerated

Participants will be in the study for about 22 weeks:

* 4 weeks for tests to see if the study might be good for them
* 12 weeks of treatment with Acthar gel
* 4 weeks to wean off Acthar gel and follow-up with the doctor

ELIGIBILITY:
Inclusion Criteria:

* Has severe or recalcitrant keratitis
* Did not respond to, or tolerate, treatment with topical cyclosporine, Lifitegrast, or any immunosuppressant to treat keratitis
* If able to reproduce, agrees to use 2 forms of effective contraception with a partner of the opposite sex for the duration of the study (through Visit 6)
* Has normal eyelids, and protocol-defined physical and medical eye attributes
* Agrees to avoid wearing contact lenses during the trial

Exclusion Criteria:

* Is pregnant or breast-feeding
* Is defined as vulnerable, or is employed by, or related to anyone involved in the study
* Has a medical condition or history that might, per protocol or in the opinion of the investigator, compromise the participant's safety or study analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (9):
- United States (9):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Global Research Management, Inc., Glendale, California
  - Eye Research Foundation, Newport Beach, California
  - Eye Care Institute, Louisville, Kentucky
  - Andover Eye Associates, Raynham, Massachusetts
  - Vita Eye Clinic, Shelby, North Carolina
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Total Eye Care, P.A., Memphis, Tennessee
  - Advancing Vision Research, LLC, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT04169061) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

REFERENCES:
- [Derived] Wirta D, McLaurin E, Ousler G, Liu J, Kacmaz RO, Grieco J. Repository Corticotropin Injection (Acthar(R) Gel) for Refractory Severe Noninfectious Keratitis: Efficacy and Safety from a Phase 4, Multicenter, Open-Label Study. Ophthalmol Ther. 2021 Dec;10(4):1077-1092. doi: 10.1007/s40123-021-00400-y. Epub 2021 Oct 20. PMID 34669183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-six participants were enrolled at 8 locations in the United States
Period: Overall Study
Arm/Group | All Participants
Started | 36
Safety Population | 36
Modified Intent to Treat (mITT) Population | 34
Completed | 31
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population
Groups:
- All Participants: Participants receive Acthar Gel administered by a shot under the skin (subcutaneous injection) per study regimen
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Improved on the Impact of Dry Eye on Everyday Life (IDEEL) Scale [Using the Symptom Bother Module at Week 12]
Description: A 12-point score reduction on the 100-point symptom bother module indicates a clinically important reduction of bothersome dry eye symptoms.
Time Frame: Week 12
Population: Participants with non-missing baseline data
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 34
Participants | 17

ADVERSE EVENTS:
Time Frame: While participating in the trial (up to 22 weeks)
Description: All serious adverse events that occurred during the trial are reported, regardless of dosing status. Non-serious treatment-emergent adverse events are included if 5% or more participants had that same event.
  Participants may have more than one event per system organ class and preferred term.
  At each level of subject summarization, a participant is counted once if the participant had one or more events.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 1/36
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 2/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=36)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=36)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT04169061/Prot_SAP_001.pdf